CLINICAL TRIAL: NCT05571397
Title: Expanding Use of Continuous Glucose Monitoring Beyond COVID in Critical Care: Impact on Nurse Work Patterns and Patient Outcomes
Brief Title: Expanding Use of CGM in Critical Care: Impact on Nurse Work Patterns and Patient Outcomes
Acronym: CGM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021H0407; G220050 (Other: FDA)
Record Dates: First submitted 2022-09-15; First posted 2022-10-07 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Intervention Model Description: CGM will be used by 100 MICU patients with glycemic control comparison with matched 100 MICU historical controls
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Dexcom CGM (Experimental): Dexcom G6
  Interventions: Device: Dexcom G6
- Historical Controls (No Intervention): Matched historical controls

INTERVENTIONS:
Device: Dexcom G6 — Continuous Glucose Monitor
  Arms: Dexcom CGM

SUMMARY:
The primary objective of this implementation study is to assess the feasibility of real time continuous glucose monitoring (CGM) implementation using a CGM plus (+) point-of-care (POC) protocol among patients on IV insulin or those with hyperglycemia (>250mg/dl) in the critical care hospital environments.

DETAILED DESCRIPTION:
This study analyzes the feasibility of inpatient real time CGM implementation through the use of a CGM + POC protocol as routine care for glycemic monitoring among patients on IV insulin or those with hyperglycemia (>250mg/dl). The investigators will examine the effects on medical intensive care (MICU) patient's (N=100) glycemic control compared to matched historical control patients (N=100) from the MICU who received fingerstick POC.

ELIGIBILITY:
Inclusion Criteria:

* adults >18 years old,
* admitted to Ohio State University Wexner Medical Center MICU and
* have hyperglycemia (glucose >250mg/dl) or are currently on IV insulin.

Exclusion Criteria:

* Current COVID-19 infection,
* Refractory shock (Levophed dose >0.5 mcg/kg/min or equivalent)
* Actively being treated for diabetic ketoacidosis (DKA)
* Actively being treated for hyperosmolar non-ketoacidosis (HONK)
* Pitting edema, anasarca, blue or purple discoloration to left upper extremity
* Treated with high dose acetaminophen (>1 gram Q6 hours)
* Treated with hydroxyurea
* Are pregnant, patients
* Using home insulin pump therapy during hospitalization, or
* Reside in a corrections institution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: EILEEN FAULDS, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexcom CGM | Historical Controls
Started | 101 | 100
Completed | 100 | 100
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexcom CGM | Historical Controls | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (15.3) | 52.7 (15.4) | 53.7 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 53 | 100
  Male | 53 | 47 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 100 | 98 | 198
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 19 | 34
  White | 83 | 77 | 160
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 200
Type of Diabetes [Count of Participants; unit: Participants]
  Type 2 Diabetes | 59 | 60 | 119
  Type 1 Diabetes | 26 | 32 | 58
  No history of diabetes | 14 | 8 | 22
  Other type of diabetes | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time in Target Glycemic Ranges
Description: Percent of time in target glycemic ranges: 100-180 mg/dl, 70-180mg/dl, 140-180mg/d
Time Frame: For duration of MICU stay which was an average of 7.6 ± 4.1 days/patient
Measure: Mean (95% Confidence Interval); unit: percentage of time in target ranges
Arm/Group | Dexcom CGM | Historical Controls
Number analyzed (Participants) | 100 | 100
percentage of time in target ranges
  70-180mg/dl | 76 [72 to 79] | 65 [61 to 69]
  100-180mg/dl | 69 [66 to 73] | 61 [56 to 64]
  140-180mg/dl | 37 [34 to 40] | 30 [27 to 33]
Statistical Analysis 1: Comparison: Dexcom CGM vs Historical Controls; Time in Range 70-180mg/dl; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dexcom CGM vs Historical Controls; Time 100-180mg/dl; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Dexcom CGM vs Historical Controls; Time 140-180mg/dl; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Percent of Time in Hypoglycemic Ranges
Description: Percent of time in hypoglycemic ranges <70mg/dl and <55mg/dl
Time Frame: For duration of MICU stay which was an average of 7.6 ± 4.1 days/patient
Measure: Mean (95% Confidence Interval); unit: Percent of time in hypoglycemic ranges
Arm/Group | Dexcom CGM | Historical Controls
Number analyzed (Participants) | 100 | 100
Percent of time in hypoglycemic ranges
  <70mg/dl | 0.41 [0.08 to 0.73] | 0.19 [0.04 to 0.34]
  <54mg/dl | 0.06 [0 to 0.16] | 0.08 [0 to 0.17]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each individual while they were enrolled in the study and wearing the continuous glucose monitor. This was an average of 7.6 ± 4.1 days.
Arm/Group | Dexcom CGM | Historical Controls
All-Cause Mortality (participants affected / at risk) | 22/100 | 23/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 8/100 | 0/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexcom CGM (N=100) | Historical Controls (N=100)
Failure to Reconsent (Investigations) | 8 (8) | 0 (0) — Subjects who were determined to be unable to provide initial consent for study enrollment were enrolled by their legally authorized representative (LAR). Per protocol, subjects are to be reconsented. Study team failed to obtain re-consent.
Failure to remove CGM when transition to hospice care (Investigations) | 2 (2) | 0 (0) — Participant study participation is to end when transition to comfort care or hospice. Study team failed to remove CGM when transitioned to hospice care

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT05571397/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT05571397/ICF_001.pdf